CLINICAL TRIAL: NCT07316712
Title: Effect of TECAR (Transfer of Energy Capacitive and Resistive) Therapy on Chronic Supraspinatus Tendinitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Ibrahem Alghamry, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005900
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Supraspinatus Tendinitis
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment + TECAR therapy (Experimental): The experimental group will receive conventional physiotherapy sessions as the active comparator group, in addition to TECAR therapy at the end of each session. Sessions will be received for three weeks (nine sessions, three times per week).
  Interventions: Other: Conventional treatment; Device: TECAR (Transfer of Energy Capacitive and Resistive) Therapy
- Conventional treatment (Active Comparator): The active comparator group will receive conventional physiotherapy sessions for three weeks (nine sessions, three times per week).
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Conventional treatment — All patients in both groups will receive conventional treatment, 3 sessions per week for 3 weeks. The conventional methods for treating supraspinatus tendinitis include shoulder swings, painless range of motion (ROM) exercises, shoulder joint active-assisted exercises, resistance exercises to improve muscle strength, and pain-reducing physiotherapy modalities like ultrasound.
Device: TECAR (Transfer of Energy Capacitive and Resistive) Therapy — Patients in the experimental group only will receive TECAR therapy, 3 sessions per week for 3 weeks. The treatment will start with an automatic capacitive energy transfer for 10 minutes. Next, the capacitive plaque will be replaced by the resistive electrode, and the neutral electrode will be fixed
  Arms: Conventional treatment + TECAR therapy

SUMMARY:
This study aims to investigate the effect of TECAR therapy on pain, shoulder range of motion, functional disability, and handgrip strength in patients with grade II supraspinatus tendinitis.

DETAILED DESCRIPTION:
Tendinopathy occurs when pain arises in a tendon near its origin or insertion due to repetitive activities and reduced functional levels. It happens when the tendon does not properly heal. Thirty percent of tendinopathies related to musculoskeletal conditions are associated with shoulder pain, and supraspinatus tendinitis is the third most prevalent problem.

The supraspinatus tendon, part of the rotator cuff of the shoulder joint, is particularly affected. Aging is also a common factor leading to supraspinatus tendon injuries. The primary function of the supraspinatus muscle is shoulder abduction, particularly during movements that elevate the arm overhead. During these motions, the supraspinatus tendon repeatedly passes beneath the acromion process of the scapula, which can result in impingement and subsequent inflammation. An unexpected force or trauma may cause a partial or complete tendon rupture if this condition progresses.

Transfer of Energy Capacitive and Resistive (TECAR) offers a unique variety of treatments for chronic and acute pathologies, with contraindications such as pregnancy, pacemakers, and sensitivity to high temperatures. It should be noted that this new technology is a valuable tool in treating various pathologies, particularly when compared with other therapies in terms of the presence and/or absence of specific positive effects. TECAR also has distinct characteristics that are effective even when other treatments fail. This therapy balances the therapist's manual skills and the specialized energy that this technology offers, resulting in increasingly satisfactory outcomes for therapists and patients.

ELIGIBILITY:
Inclusion Criteria:

* Supraspinatus Tendinitis grade II based on Neer's classification, confirmed by special tests, signs, and symptoms of grade I and II Supraspinatus Tendinitis for the past month, and taking non-steroidal anti-inflammatory drugs as suggested by the physician.
* All patients will have a body mass index between 18.5 and 29.9 kg/m².

Exclusion Criteria:

* Other grades of Supraspinatus Tendinitis.
* Any past shoulder surgical interventions.
* Instability of the shoulder joint due to other reasons, Acromioclavicular Joint Arthritis.
* Non-cooperative subjects.
* Diabetes
* Pregnant or lactating women.
* Serious neuromuscular or cardiovascular diseases.
* Systemic illness and severe COVID-19 cases will be excluded from this study.
* Pacemakers
* Heat Sensitivity
* Metal Implants

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain Intensity of Shoulder Joint by Numerical Rating Scale (NRS) | 3 weeks
  The Numerical Rating Scale (NRS) will evaluate shoulder pain when using the NRS. Patients will be asked to rate their pain on a scale from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain possible.

SECONDARY OUTCOMES:
Assessment of Shoulder abduction range of motion | 3 weeks
  A digital goniometer will be used to assess shoulder joint abduction range of motion in patients with chronic supraspinatus tendinitis before and after the treatment sessions. Measurements will be taken with the patient in the supine position. The fulcrum of the goniometer will be centered at the anterior aspect of the acromion process, the stationary arm will be aligned parallel to the midline of the torso, and the moving arm will be aligned with the midline of the humerus, pointing toward the medial epicondyle of the elbow.
Assessment of Shoulder External Rotation range of motion | 3 weeks
  Shoulder joint external rotation range of motion will also be assessed using a digital goniometer before and after the treatment sessions in patients with chronic supraspinatus tendinitis. The patient will be positioned supine during measurement. The fulcrum of the goniometer will be centered over the olecranon process of the elbow, the stationary arm will be aligned perpendicular to the floor, and the moving arm will be aligned with the ulna, pointing toward the ulnar styloid process.
Assessment of Handgrip strength by handheld dynamometer | 3 weeks
  A JAMAR hand dynamometer (Sammons Preston Inc, Bolingbrook, IL, USA) will be used to measure grip strength in kilograms. The Jamar is small and portable but relatively heavy at 1.5 lb. The dial reads force in both kilograms and pounds, with markings at intervals of 2 kg or 5 lb, allowing assessment to the nearest 1 kg or 2.5 lb. The reading error is reported to be greater at lower loadings. This method has high test-retest reliability. Also, it has both inter and intra-rater reliability.
Assessment of Functional disability by QuickDASH Scale (Arabic Version) | 3 weeks
  The QuickDASH includes 30 items, with six items about symptoms (3 about pain, 1 for tingling/numbness, 1 for weakness, 1 for stiffness) and 24 about function (21 about physical function, 3 about social/role function). For each question, the subject rated the performance in the last week on a 5-point scale (1 = no difficulty to perform or no impact; 5 = unable to do or high impact). The raw score is the sum of all answers (maximum score: 150; minimum score: 30). The raw score is transformed into a zero to 100 scale (= total DASH). Zero is no disability and 100 maximum disability.

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa Kenawy Atta, PhD, Study Chair — Assistant Professor, Cairo University; Hend Hamdy Mohamed Ahmed, PhD, Study Director — Lecturer, Cairo university
Locations (1):
- CAN Center outpatient clinic, Cairo, Egypt